CLINICAL TRIAL: NCT07052721
Title: A Randomized, Single-Blinded, Sham-Controlled Study Evaluating the Efficacy and Safety of RELAY, a Device Enabling Both Local Anesthetic Delivery and Neuromodulation Following Shoulder or Foot Surgery
Brief Title: Randomized Study of an Analgesic Device Enabling Local Anesthetic Delivery and Neuromodulation After Shoulder/Foot Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Gate Science (Industry)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RELAY Randomized
Record Dates: First submitted 2025-06-28; First posted 2025-07-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Tears; Shoulder Injuries; Hallux Valgus; Ankle Arthropathy; Clavicle Fracture
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Injuries; Hallux Valgus

STUDY DESIGN:
Intervention Model Description: Single center, randomized, observer- and participant-masked, sham-controlled parallel group study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Pulse generators are available that are capable of either (1) passing electrical current; or (2) not passing electrical current. Importantly, these 2 modes (active and sham) are indistinguishable in appearance, and therefore investigators, participants, and all clinical staff will be masked to treatment group assignment, with the only exception being the unmasked individuals who insert the RELAY and program the stimulator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active Neuromodulation (Experimental): RELAY catheter will be inserted under ultrasound guidance followed by a local anesthetic bolus injection. If a patient's surgeon requests a postoperative continuous peripheral nerve block, a ropivacaine 0.2% infusion will be initiated in the recovery room. Within the recovery room, the stimulators will be connected to participants' phones and turned on. The catheters will be removed on postoperative day 7.
  Interventions: Device: Experimental Treatment
- Sham Neuromodulation (Sham Comparator): RELAY catheter will be inserted under ultrasound guidance followed by a local anesthetic bolus injection. If a patient's surgeon requests a postoperative continuous peripheral nerve block, a ropivacaine 0.2% infusion will be initiated in the recovery room. Within the recovery room, the stimulators will be connected to participants' phones and turned on, but no current will reach the electrodes or patient's body. The catheters will be removed on postoperative day 7.
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: Experimental Treatment — Percutaneous peripheral nerve stimulation with a frequency of 100 Hz, a pulse duration of 100 µs, and a current amplitude of 0.001-10 mA (1-10,000 µA). Participants will adjust the amplitude, as needed.
  Other Names: percutaneous peripheral nerve stimulation
  Arms: Active Neuromodulation
Device: Sham Comparator — SHAM percutaneous peripheral nerve stimulation with a frequency of 100 Hz, a pulse duration of 100 µs, and a current amplitude of 0.001-10 mA (1-10,000 µA). Participants can adjust the amplitude, as needed; but no electrical current will ever reach the patient's body.
  Other Names: Placebo
  Arms: Sham Neuromodulation

SUMMARY:
Postoperative pain remains undertreated with inadequate analgesic options. Opioids have well-known limitations for both individuals and society; single-injection and continuous peripheral nerve blocks provide intense analgesia but are limited in duration to 24-72 hours; and current neuromodulation options-with a duration measured in weeks and not hours-are prohibitively expensive and require an additional procedure. One possible solution is a device currently under investigation to treat postoperative pain. The RELAY system (Gate Science, Moultonborough, New Hampshire) is comprised of a basic catheter-over-needle device to allow administration of a single-injection of local anesthetic via the needle (or catheter) followed by a perineural local anesthetic infusion via the remaining catheter (when desired). Subsequent to the local anesthetic administration, instead of removing the catheter as with all previous continuous peripheral nerve block equipment, electric current may be delivered via the same catheter and an integrated pulse generator for up to 28 days. This is potentially revolutionary because it would allow an anesthesiologist to deliver (1) a single-injection peripheral nerve block; (2) a continuous peripheral nerve block; and (3) neuromodulation using a single device that can theoretically be placed in the same amount of time required for a single-injection peripheral nerve block. Instead of providing fewer than 24 hours of postoperative analgesia, up to 28 days of pain control could be delivered without disruption of existing practice patterns. The ultimate objective of the proposed investigation is to investigate the post-operative analgesic potential of this investigational device and prepare for a pivotal multicenter clinical trial.

DETAILED DESCRIPTION:
For individuals of childbearing potential, a sample of urine will be collected before any study interventions to confirm a non-pregnant state (this is standard procedure for all surgical patients). Participants will have standard external monitors placed and oxygen delivered by facemask or nasal cannula. The peripheral nerve block site(s) will be cleansed with chlorhexidine gluconate and isopropyl alcohol. Intravenous sedation/analgesia with midazolam and/or fentanyl will be titrated for patient comfort as is standard for peripheral nerve block administration. The nerves treated will include the sciatic proximal to the popliteal crease for foot surgery and the brachial plexus for shoulder/clavicle surgery. The target nerve(s) will be visualized with ultrasound using a transverse cross-sectional (short axis) view and a skin wheal of local anesthetic will be raised inferior to the transducer to anesthetize the skin and then the track towards the target.

Participants will be randomly allocated to one of two possible treatments groups: (1) Neuromodulation or (2) Sham [Control].

Randomization will be stratified by anatomic location (shoulder and foot/ankle surgery) in a 1:1 ratio and in blocks of 2. Computer-generated randomization lists will be created by the UC San Diego Investigational Drug Service and participants allocated to the treatment groups in sequential order. Pulse generators are available that are capable of either (1) passing electrical current; or (2) not passing electrical current. Importantly, these 2 modes (active and sham) are indistinguishable in appearance, and therefore investigators, participants, and all clinical staff will be masked to treatment group assignment, with the only exception being the unmasked individuals who insert the RELAY and program the stimulator.

The RELAY system with the integrated needle will be inserted adjacent to the target nerve with an in-plane approach. Dextrose 5% in water (1-20 mL) will be injected via the needle to open a space around the target nerve(s), the catheter advanced, and the needle subsequently withdrawn.

Active treatment group. For participants randomized to active treatment, electrical current will be introduced with increasing intensity using the most proximal and distal electrodes (control provided by the Gate Keeper app from an investigator's phone or tablet). Accurate lead placement will be confirmed with subject reports of comfortable sensations over the surgical site without eliciting muscle contractions. The minimum threshold and maximum comfortable amplitudes will be determined along with the optimal frequency, pulse duration, and anode/cathode. Starting from the lowest possible current the investigators increase the current until the participant states that they feel a "buzzing" sensation (some describe it as a "comfortable massage"). That is the minimal sensed current. The investigators will then continue increasing with the instructions to let them know when it starts to be less comfortable-and to stop us before it hurts. That is the maximum comfortable current. The stimulator will be then set to deliver the minimum threshold amplitude and turned off for surgery.

Sham treatment group. For participants receiving sham treatment, electric current will not reach the electrodes, but the investigators will connect to the RELAY to the mobile phone or tablet just as with the active group and set the parameters as follows: anode (distal), cathode (proximal), frequency (100 Hz), pulse duration (100 µs), and amplitude (5 mA).

Local anesthetic for active and sham groups. Local anesthetic (10 mL of lidocaine 2% with epinephrine) will be injected with negative aspiration every 3 mL and resulting sensory block confirmed to ensure accurate catheter tip placement. Following block confirmation (sensory deficits in the expected nerve distributions), the RELAY will be affixed with both surgical adhesive (2-Octyl 2-cyanoacrylate) at the entry site and a chlorohexidine-impregnated occlusive dressing. Subsequently, 10 mL of bupivacaine 0.5% with epinephrine will be injected negative aspiration every 3 mL along with a supplemental single-injection saphenous nerve block for foot/ankle surgery.

Intraoperatively, surgeons will be permitted to infiltrate the surgical area with long-acting local anesthetic as their common practice dictates.

Postoperatively, the stimulators will be connected to participants' phones and turned on.

If a patient's surgeon requests a postoperative continuous peripheral nerve block, a ropivacaine 0.2% infusion will be provided per standard UC San Diego protocol using a 200 mL reservoir. This will provide an infusion lasting through postoperative day 1, and is approximately 1 day shorter than is our current standard practice.

After 7 days, participants in both the active and sham groups, themselves or their caretaker will remove the occlusive dressing and withdraw the catheter (and integrated electrodes) with gentle traction and rotation at home. The devices are single-use and disposable.

Following study completion, the results will be mailed electronically or by the United States Postal Service to all enrolled participants in written form using non-technical (e.g., "layperson") language.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants of at least 18 years of age
2. Undergoing a rotator cuff repair, total shoulder arthroplasty, clavicle fracture ORIF, or foot/ankle surgery anticipated to have moderate-to-severe pain for a week after surgery (e.g., ankle arthroplasty/arthrodesis)
3. At least a single-injection peripheral nerve block(s) planned
4. An Android or Apple smartphone able to download the Gate Keeper controller app

Exclusion criteria:

1. Chronic opioid or tramadol use (daily within prior 2 weeks and duration > 4 weeks)
2. Neuro-muscular deficit of the surgical limb
3. Compromised immune system based on medical history (e.g., immunosuppressive therapies such as chemotherapy, radiation, sepsis, infection), or other conditions that places the subject at increased risk of infection
4. Implanted spinal cord stimulator, cardiac pacemaker/defibrillator, deep brain stimulator, or other implantable neurostimulator whose stimulus current pathway may overlap
5. History of bleeding disorder
6. Antiplatelet or anticoagulation therapies other than aspirin
7. Allergy to skin-contact materials (occlusive dressings, bandages, tape etc.)
8. Incarceration
9. Pregnancy
10. Moderate pain (NRS > 3) in an anatomic location other than the surgical site
11. Anxiety disorder
12. History of substance misuse
13. Inability to communicate with the investigators
14. Inability to contact the investigators during the treatment period, and vice versa (e.g., lack of telephone access)
15. Allergy to amide local anesthetics
16. Morbid obesity (body mass index > 40 kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Average daily pain intensity postoperative days 1-7 | Days 1-4 and 7
  The median of 4 daily "average" pain intensity scores for Days 1-4 and 7 as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst) collected on Days 2, 3, 4, and 7 for the previous 24 hours each.

SECONDARY OUTCOMES:
Cumulative opioid use 1st week | The first 7 days following surgery
  The cumulative opioid use measured in oxycodone equivalents during the first 7 days following surgery
Brief Pain Inventory (interference sub scale) | Postoperative days 3 and 7
  The Brief pain Inventory (short form) is an instrument specifically designed to assess pain and its impact on physical and emotional functioning. The brief Inventory is comprised of three domains: (1) pain, with four questions involving "worst", "average" and "current" pain levels using a 0-10 numeric rating scale;(2) percentage of relief provided by pain treatments with one question [reported score is the percentage divided by 10 and then subtracted from 10: 0=complete relief,10=no relief] and, (3) interference with 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference;10=complete interference]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. This outcome will include the interference subscale.
Worst/maximum daily pain intensity postoperative days 2-7 | Days 1-4 and 7
  The median of 4 daily "worst" pain intensity scores for Days 1-4 and 7 as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst) collected on Days 2, 3, 4, and 7 for the previous 24 hours each.
Awakenings due to pain 1st week, cumulative | Collected on postoperative days 1-7
  Cumulative number of nightly awakenings due to pain
Nightly awakenings due to pain | Collected on postoperative days 1-4, 7, 8, and 14
  Number of awakenings due to pain each night
Daily "average" pain intensity | Postoperative Days 1-4, 7, 8, and 14
  The "average" pain intensity score on each postoperative day as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst)
Daily "worst" pain intensity | Postoperative Days 1-4, 7, 8, and 14
  The "worst" pain intensity score on each postoperative day as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst)
Daily oxycodone consumption | Postoperative Days 1-4, 7, 8, and 14
  The cumulative opioid use from the previous 24 hours measured in oxycodone equivalents collected on Days 1-4, 7, 8, and 14
Percentage of group avoiding severe pain (NRS>6) | Postoperative Days 1-14
  Percentage of each treatment group which never reported a worst pain score > 6 as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst) following recovery room discharge
Percentage of group avoiding opioids | Postoperative Days 1-14
  Percentage of each treatment group which never used opioids following recovery room discharge
Day of discharge | Postoperative Days 0-14
  The postoperative day that the patient is discharged home or to a skilled nursing facility
Blinding assessment | Postoperative Day 7
  Patients are asked if they think they received active treatment, sham treatment, or are not sure of which treatment they received

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided